CLINICAL TRIAL: NCT03941340
Title: A Phase I Mass Balance and Biotransformation Study of Orally Administered [14C]-Alflutinib Mesylate (AST2818) in Chinese Healthy Male Volunteers
Brief Title: Study Evaluating the Mass Balance And Biotransformation of Single Dose[14C] AST2818 in Chinese Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allist Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20190130
Record Dates: First submitted 2019-04-24; First posted 2019-05-07 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Healthy Male Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]-AST2818 80mg (oral solution) (Experimental): Volunteers will receive 80 mg [14C]-AST2818 containing a nominal 100 μCi activity, administered by mouth, as a solution.
  Interventions: Drug: [14]-AST2818

INTERVENTIONS:
Drug: [14]-AST2818 — Volunteer will receive a single oral dose of 80 mg /100 u Ci [14C]-AST2818 as a solution on Day 1

SUMMARY:
Study to Evaluate the Mass Balance and Biotransformation of Single Dose[14C] AST2818 in Chinese Healthy Male Volunteers

DETAILED DESCRIPTION:
A Phase I Mass Balance and Biotransformation Study of Orally Administered [14C]-Alflutinib Mesylate (AST2818) in Chinese Healthy Male Volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult;
2. Body weight: The body mass index varies in the range of 19 - 26 kg/m2 (including 19 and 26 kg/m2);
3. Signing the informed consent forms by oneself ;
4. Be able to communicate well with the researcher and be able to complete the trial in accordance with the program.

Exclusion Criteria:

1. Those with abnormal examination and clinical significance ( including Physical examination, routine laboratory examination (blood routine, urine routine, fecal routine + Occult blood, blood biochemistry, blood coagulation routine, thyroid function), 12-lead electrocardiogram, X-ray (positive position), abdominal B-mode ultrasonography (liver, gallbladder, pancreas, spleen and kidney), etc)；
2. Those with routine urine examination showed positive urinary protein；
3. Those with QTcF > 470 msec in resting state, corrected by ECG during screening period；
4. Those with HBsAg , HBeAg and HCVAb were positive；
5. Those with HIVAb was positive；
6. Those with treponema pallidum Ab was positive；
7. Those who take any drugs that inhibit or induce the CYP450 enzyme (i.e., inducers- barbiturates, tegretol, phenytoin, rifampicin, hexadecadrol, rifabutin, rifapentini; inhibitors- SSRI-antidepressant, cimetidine, diltiazem, macrolides, verapamil, imidazoles- antifungal drugs) 30 days prior to screening period；
8. Those who take any drug, health care products (including vitamins), chinese traditional medicine 14 days prior to screening period；
9. Those who participated other clinical trials or took the investigational drug 3 months prior to screening period, or prepare to take part in other clinical trials within 1 month after finishing this trial；
10. Those who have history of organic heart disease, heart failure, myocardial infarction, angina, unexplained arrhythmia, torsional ventricular tachycardia, ventricular tachycardia and QT prolonged syndrome, or have the family history (Genetic proof or a close relative of sudden cardiac death at a young age) and symptom of QT prolonged syndrome ；
11. Those who have severe disease of ophthalmic system, e.g., corneal, conjunctiva and eyelid diseases;
12. Those who have undergone major surgery within the first 6 months of the screening period or have no complete surgical incision; major procedures include, but are not limited to, any operator with significant bleeding risk, prolonged general anesthesia, or incisional biopsy or significant traumatic injury;
13. Those who have but not limited to circulatory system, endocrine system, nervous system, digestive system, urinary system, or have the history of blood, immunity spirit and metabolism diseases；
14. Those who have allergic constitution, including being definitely allergic to TKIs or any ingredients of this trial drugs，any food materials or have special demands for foods，and cannot comply with the rule of unified diet；
15. Those who have history of hand and foot syndrome；
16. Those who have haemorrhoids or perianal disease with regular/ongoing hematochezia；
17. Those who have coagulation dysfunction or other diseases of the blood system;
18. Those who have history of tumor；
19. Those who have habitual constipation or diarrhea, irritable bowel syndrome, inflammatory bowel disease；
20. Those who have history of alcohol abuse (it was defined as that the daily alcohol consumption was higher than the following criteria: the weekly alcohol consumption was higher than 14 units of alcohol (1 unit= 360 ml beers/45 ml liquor containing 40% alcohol/150ml grape wine) 6 months prior to screening period, or the alcohol breath test results ≥20 mg/dl during screening period；
21. Those who smoked daily >5 sticks of cigarette 3 months prior to first dose or cannot give up smoking during study；
22. Those have history of drug abuse or taking soft drug (i.e., marihuana) 3 months prior to screening period or taking hard drugs (i.e., cocaine, amphetamines, benzodiazepine, etc.); or the results of urine test in drugs were positive;
23. Those who were used to drink grapefruit juice or overconsumption of tea, coffee, and the drink with caffeine; and cannot give up them during test；
24. Those who need long-term exposure to radiation, or who have been exposed to significant radiation (> 2 chest/abdominal CT scans or more than 3 other X-ray scans) or who have participated in the labeling test of radiopharmaceuticals within one year before the test;
25. Those who have fertility planning within the range of starting trial - 1 year after finishing trial, or disagree with the regulation and their mate should take strict contraception (taking condoms, contraceptive sponges, contraceptive gels, contraceptive membranes, intrauterine devices, oral or injectable contraceptives and subcutaneous implants, etc.)；
26. Those who have excessive bleeding or blood donation (400ml) 3 months prior to screening period, or planned to donate blood 1 month after finishing this trial；
27. Those who cannot complete this study because of other reasons, or any factors judged by investigator that the participants cannot meet.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
The distribution of AST2818 in the whole blood and plasma and whole radioactive pharmacokinetics following the single orally administered [14C]-AST2818 in healthy male volunteers. | Blood samples (hrs) - 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, every 24 to 504, 672, 840, 1008, 1176, 1344, 1512, 1680, 1848 and 2016.
  The percentage of radioactive dose of [14C] radiolabelled AST2818 recovered in blood and in total, up to Day 85（p.s:The administration time on the first day is 7:30 am）
Quantitive analysis of whole radioactivity of excrement of orally administered [14C]-AST2818 in healthy volunteers to obtain the mass balance data and the main excretion pathway in human body. | Urine and faeces (hrs): 0-4, 4-8, 8-12, 12-24, every 24 to 504, 624-672, 792-840, 960-1008, 1128-1176, 1296-1344, 1464-1512, 1632-1680, 1800-1848 and 1968-2016.
  The percentage of radioactive dose of [14C] radiolabelled AST2818 recovered in urine, faeces and in total, up to Day 85（p.s:The administration time on the first day is 7:30 am）
Quantitive analysis of the concentrations of AST2818 and AST5902 (Metabolite of AST2818) in plasma using the validated LC-MS/MS to obtain pharmacokinetic data; | Blood samples (hrs) - 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, every 24 to 504, 672, 840, 1008, 1176, 1344, 1512, 1680, 1848 and 2016.
  The concentrations of AST2818 and AST5902 in plasma up to Day 85（p.s:The administration time on the first day is 7:30 am）
Proportion of different metabolites in healthy volunteers after oral administration of [14C]-AST2818 | Blood samples (hrs) - 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, every 24 to 504, 672, 840, 1008, 1176, 1344, 1512, 1680, 1848 and 2016.
  Proportion of different metabolites
Types of adverse events assessed by CTCAE v5.0 that occurred during the trial | Baseline (Day-1) to Day 85（p.s:The administration time on the first day is 7:30 am）
  Types of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: LiYan Miu, Principal Investigator — First Affiliated Hospital of Soochow University
Locations (1):
- First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China